CLINICAL TRIAL: NCT06420947
Title: Application of Electrically Driven Atomized Surface Anesthesia to Awake Endotracheal Intubation in Patients With Predictably Difficult Airway.
Brief Title: Application of Electrically Driven Atomized Surface Anesthesia in ATI in Patients With Predictably Difficult Airway.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Henan xixi
Record Dates: First submitted 2024-05-12; First posted 2024-05-20 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia, Endotracheal
Keywords: Lidocaine atomized particles; Nebulization; Awake tracheal intubation; Individual topicalization technique
MeSH Terms: interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Experimental): Participants in the A group received 2% lidocaine by A model atomizer.
  Interventions: Other: atomizer
- Group B (Experimental): Participants in the B group received 2% lidocaine by B model atomizer.
  Interventions: Other: atomizer
- Group C (Experimental): Participants in the C group received 2% lidocaine by C model atomizer.
  Interventions: Other: atomizer
- Group D (Experimental): Participants in the D group received 2% lidocaine by D model atomizer.
  Interventions: Other: atomizer

INTERVENTIONS:
Other: atomizer — Participants received 2% lidocaine by atomizer.
  Other Names: a wearable and disposable vibrating mesh nebulizer

SUMMARY:
This is a parallel and randomized-controlled clinical study aimed to identify the optimized size of atomized particles of 2% lidocaine that can provide the best topical anesthesia during ATI. To determine the effect of nebulization with different sizes of atomized particles of 2% lidocaine on cough, reaction, and comfort during ATI in patients with predicted difficult airway.

ELIGIBILITY:
Inclusion Criteria:

Patients with distinctly difficult airways：(1) Patients with medical history indicating difficult airways.(2) Patients suffering from severe burn scars.(3) Patients suffering from severe obstructive sleep apnea syndrome.(4)Patients suffering from severe congenital dysplasia.

Patients with suspected difficult airway:

Patients with risk factors underwent a medical history for evaluation:(1)Patients with ankylosing spondylitis.(2) Patients with rheumatoid arthritis.(3)Patients with degenerative osteoarthritis.(4)Patients with epiglottitis. (5)Patients with acromegaly.(6)Patients with morbid obesity.(7)Patients with subglottic stenosis. (8) Patients with enlarged thyroid or tonsils.(9)Patients with mediastinal mass.(10)Patients with throat tumors.

Patients with risk factors underwent a physical examination for evaluation:(1)Patients with BMI > 26 kg/m2. (2)Patients with Mallampati class 3 or 4. (3)Patients with thyromental distance<60 mm (corresponding to an average distance of 3 finger breadths).(4)Patients with limited mouth opening with interincisor distance<30 mm.(5)edentulous patients.(6)When the patient closed his mouth in a natural state, the upper incisor was situated in front of the lower incisor.(7)When the mandible is extended forward, the lower incisors of the patient can not protrude beyond the upper incisors.(8)The patient's jaw exhibits stiffness, with minimal elasticity or presence of a tumor.(9)The patients have a short neck with a thick circumference.(10)The patients are unable to touch their chest wall with their jaw, or extend their neck.(11)The patients's palate shape is either characterized by a high arch or is extremely narrow.

Exclusion Criteria:(1) refusal to participate in the study; (2) airway bleeding; and (3) known allergies to local anesthetics.

-

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
cough score | during intubation
  Investigators will record cough score during intubation.

SECONDARY OUTCOMES:
reaction and discomfort scores | during intubation.
  Investigators will record reaction and discomfort scores during intubation.
intraoperative hemodynamic parameters | endotracheal tube insertion, inflation of the tracheal tube cuff and 1 minute after endotracheal tube insertion
  endotracheal tube insertion inflation of the tracheal tube cuff systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR)

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqiang Zhang, PHD, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Li C, Sun M, Zhang L, Wang G, Lu J, Xie Z, Zhang J. Nebulization with differently sized 2% lidocaine atomized particles in awake tracheal intubation by video laryngoscopy: a proof-of-concept randomized trial. BMC Anesthesiol. 2025 Jul 1;25(1):321. doi: 10.1186/s12871-025-03178-9. PMID 40596861